CLINICAL TRIAL: NCT03723304
Title: The Intention-to-treat Effect of Bridging Therapies in the Setting of Milan-in Patients Waiting for Liver Transplantation
Brief Title: The Intention-to-treat Effect of Bridge Therapies in the Setting of Milan-in Patients
Status: Completed | Type: Observational
Sponsor: European Hepatocellular Cancer Liver Transplant Group (Other)
Responsible Party: Sponsor
Other Study IDs: #0002
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Liver Cancer; Transplant; Failure, Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct liver transplant: All the cases listed for liver transplantation and then transplanted/dropped-out without undergoing any neo-adjuvant loco-regional treatment
  Interventions: Procedure: Direct liver transplant
- Bridging followed by transplant: All the cases listed for liver transplantation and then transplanted/dropped-out after undergoing at least one neo-adjuvant loco-regional treatment
  Interventions: Procedure: Bridging followed by transplant

INTERVENTIONS:
Procedure: Bridging followed by transplant — Trans-arterial chemoembolization or percutaneous alcohol injection or radio-frequency ablation during the waiting time followed by liver transplant
  Groups: Bridging followed by transplant
Procedure: Direct liver transplant — Direct liver transplant (no neoadjuvant approaches during the waiting time period)
  Groups: Direct liver transplant

SUMMARY:
In patients with hepatocellular cancer (HCC) meeting the Milan Criteria (MC), the usefulness of loco-regional therapies (LRT) in the context of liver transplantation (LT) is still debated. The inconsistent literature data are the result of initial selection biases among treated and untreated patients. In order to overcome these shortcomings, an inverse probability of treatment weighting (IPTW) analysis was done in a large patient cohort. After using a competing-risk analysis, the primary end-point of the study aims at identifying the risk factors of HCC-specific LT failure, defined as pre-LT tumour-related drop-out or post-LT recurrence.

DETAILED DESCRIPTION:
Liver transplantation (LT) is the best curative treatment of hepatocellular cancer (HCC) developed in an underlying liver disease. LT is considered as an oncologic successful procedure when a long-term post-transplant tumour-free survival is obtained. Conversely, a failure is equal to pre-transplant drop-out, post-transplant tumour recurrence or death. Due to the allograft scarcity, a HCC patient waiting for a LT is most often treated using neo-adjuvant loco-regional therapies (LRT) in order to minimise the risk of drop-out. When the tumour burden meets the Milan Criteria (MC) at moment of diagnosis, such an approach is called "bridging towards LT".

Two recent international guidelines underlined the importance of the bridging strategy, due to its potential to reduce the risk of pre-LT drop-out and post-LT recurrence. This is especially valid in the case in which a partial/complete tumour response is achieved before LT. Unfortunately, the quality of the evidence obtained from the currently available literature is low due to the lack of randomized controlled trials (RCT). Actually, it is inconceivable to realize RCT in this setting because of logistical and, even more, ethical reasons. Consequently, the majority of reported studies just compare post-LT outcome of treated and untreated patients, failing thereby to analyse the clinical course from an intention-to-treat (ITT) point of view.

Even when looking at studies including the waiting list period, one should keep in mind that substantial differences may exist among initially bridged vs untreated HCC patients regarding tumour burden. In order to overcome these limits, a retrospective analysis of a large European population of MC-IN HCC patients listed for LT was done. After "balancing" this cohort with an inverse probability of treatment weighting (IPTW), we investigated the risk factors for tumour-specific LT failure, especially focusing at the role of LRT.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18-year old) listed for liver transplant with a morphologic and/or histologic confirmed hepatocellular cancer

Exclusion Criteria:

* Milan Criteria-out status at first referral
* transplantation or de-listing before January 1, 2001
* other means of loco-regional treatments such as partial hepatectomy, trans-arterial radio-embolization or external radiotherapy
* misdiagnosed mixed hepatocellular-cholangiocellular cancer or cholangiocellular cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological/post-bioptic diagnosis of hepatocellular cancer listed for liver transplantation receiving or not receiving any neo-adjuvant treatment before transplant/drop-out
Sampling Method: Probability Sample
Enrollment: 1083 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Tumour-specific liver transplant failure rate | up to 5 years from first referral
  Any case of tumor-related drop-out during the waiting list period or post-transplant recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Quirino Lai, MD PhD, Principal Investigator — UCL Brussels
Locations (1):
- UCL, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai Q, Vitale A, Iesari S, Finkenstedt A, Mennini G, Onali S, Hoppe-Lotichius M, Manzia TM, Nicolini D, Avolio AW, Mrzljak A, Kocman B, Agnes S, Vivarelli M, Tisone G, Otto G, Tsochatzis E, Rossi M, Viveiros A, Ciccarelli O, Cillo U, Lerut J; European Hepatocellular Cancer Liver Transplant Study Group. The Intention-to-Treat Effect of Bridging Treatments in the Setting of Milan Criteria-In Patients Waiting for Liver Transplantation. Liver Transpl. 2019 Jul;25(7):1023-1033. doi: 10.1002/lt.25492. PMID 31087772